CLINICAL TRIAL: NCT07016321
Title: Emetine for Viral Outbreaks: A Phase 2/3 Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Emetine for Dengue Fever (a.k.a. EVOLVE Antiviral Initiative)
Brief Title: Emetine for Viral Outbreaks (a.k.a. EVOLVE Antiviral Initiative)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Bharatpur Hospital Chitwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00486563
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Emetine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three arms: intervention arm #1 (6 mg emetine), intervention arm #2 (12 mg emetine), or the control arm (matching oral placebo) based on a pre-designed scheme of block randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Emetine 6 mg (Active Comparator): Participants take 6mg Emetine pill for 10 consecutive days
  Interventions: Drug: Emetine Hydrochloride 6mg
- Emetine 12 mg (Active Comparator): Participants take 12mg Emetine pill for 10 consecutive days
  Interventions: Drug: Emetine Hydrochloride 12mg
- Placebo (Placebo Comparator): Participant take a placebo for 10 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emetine Hydrochloride 6mg — To administer Emetine Hydrochloride 6mg orally for 10 consecutive days to evaluate the efficacy and safety of emetine for symptomatic dengue patients.
  Arms: Emetine 6 mg
Drug: Placebo — Participant take a placebo for 10 consecutive days.
  Arms: Placebo
Drug: Emetine Hydrochloride 12mg — To administer Emetine Hydrochloride 12mg orally for 10 consecutive days to evaluate the efficacy and safety of emetine for symptomatic dengue patients.
  Arms: Emetine 12 mg

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of emetine administered orally for symptomatic patients aged 18-65 years infected with the dengue virus. The main questions it aims to answer are:

1. Does emetine reduce 28-day mortality or progression to severe dengue (severe plasma leakage, severe bleeding, or severe organ involvement)?
2. What are the safety outcomes of emetine, including serious adverse events and toxicities?

Participants will be asked to:

1. Take either 6mg emetine, 12mg emetine, or a placebo pill for 7 consecutive days as part of the treatment regimen.
2. Have blood samples taken for at least 5 days to monitor viral load, inflammatory markers, and safety parameters.
3. Be monitored by healthcare staff for daily vital signs and symptoms for clinical assessments for 28 days.

DETAILED DESCRIPTION:
Dengue fever is a mosquito-borne viral infection caused by the dengue virus (DENV), which belongs to the Flaviviridae family. It is transmitted primarily by Aedes aegypti and Aedes albopictus mosquitoes. Dengue is recognized as one of the top ten global public health threats, affecting an estimated 390 million people annually, with approximately 96 million cases manifesting clinically. Globally, dengue has seen a significant rise in incidence, with a 30-fold increase in the past 50 years. There is currently no antiviral agent proven to work against it. Dengue fever is endemic in Nepal with cyclical outbreaks. The country relies on supportive treatment. This often includes intravenous fluids and, in rare cases, steroids and organ support. Effective antiviral agents could significantly reduce the burden of dengue by preventing disease progression and reducing transmission.

In vitro and in vivo studies have suggested strong antiviral activity of emetine against SARS-CoV-2, dengue, Ebola, cytomegalovirus, and several other viruses. Low et al. had carefully demonstrated that emetine inhibited all four serotypes of DENV infection in cell lines by inhibiting the viral RNA synthesis or the viral protein translation pathway. In the past, emetine, an alkaloid extracted from ipecacuanha roots, has been widely used in the human treatment of amoebic dysentery, amoebic liver abscess, and several viruses such as herpes simplex, herpes zoster, influenza, hepatitis, and mumps. Because of cardiotoxicity (cardiac dysrhythmias), emetine was replaced by metronidazole. The toxicity was unequivocally associated with high-dose emetine (60 mg/day for 10 days to achieve an minimum inhibitory concentration (MIC) of 25 micromol (µM) against Entamoeba histolytica; however, the cardiovascular side-effects were minimal or none when emetine was used for various indications in low dose (<20 mg/day). The investigators have recently shown that by lowering the standard amoebicidal dose by a factor of 10, emetine can inhibit viral replication while avoiding cardiovascular toxicity.

Phase 1 and 2 studies have been previously carried out. The investigators' clinical trial to evaluate emetine against SARS-CoV-2 is currently approved by Johns Hopkins Medicine (JHM) Institutional Review Board (IRB) (IRB00283778) and is ongoing in Nepal. The investigators have enrolled a few patients in this trial and have not encountered any toxicity. Given the broad-spectrum antiviral activity of emetine, the investigators now plan to evaluate emetine's efficacy and safety in the treatment of symptomatic dengue fever in a clinical trial. The investigators hypothesize that emetine will be efficacious against dengue at low doses. By evaluating its efficacy against dengue, this research can directly inform treatment strategies for patients in over 100 countries, since about 50% of the global population is at risk of dengue fever. In the past, emetine was an essential World Health Organization (WHO)- and FDA-approved drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Admitted to the hospital
3. Laboratory-confirmed infection with dengue virus within the last 5 days and preferably within the last 3 days. Testing for dengue virus using positive Nonstructural protein 1(NS1) strip assay or reverse-transcriptase polymerase chain reaction (RT-PCR)
4. Having two or more clinical symptoms (fever, headache, retro-orbital pain, myalgia, arthralgia, rash, hemorrhagic manifestations, or leucopenia, gastrointestinal symptoms) with the onset of fever within 72 hours of presentation, and
5. Able to provide voluntary informed consent and comply with all study procedures and visits.

Exclusion Criteria:

1. Age ≥65 years
2. Pregnant or breastfeeding
3. Current or recent use of the study drug
4. Known allergy to study drug
5. Current or planned participation in another pharmacological interventional trial in the next 10 days
6. Participants with known past history of dengue infection
7. Participants on aspirin, anticoagulants, or with other conditions that might increase the risk of bleeding
8. Participants on immunosuppressive agents, including long-term steroids
9. Severe dengue as defined by the WHO 2009 revised case classification.
10. Individuals with long-term immunosuppressive agents such as anti-cancer chemotherapy or radiation therapy within the past 6 months, or those on systemic corticosteroid therapy
11. History of prior vaccination against dengue fever within one year.
12. Patients who have recently used ayurvedic or herbal medications for dengue or any other conditions in the last 7 days (eg, Papaya leaf extract)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate effectiveness of emetine in dengue patients assessed by 28-day mortality or progression | 28 days
  28-day mortality or progression to severe dengue, defined as severe plasma leakage, severe bleeding, or severe organ involvement (death and severe dengue will be assessed as a composite outcome)
Safety of emetine assessed by number of adverse events | Up to 28 days
  Record serious adverse events and toxicities by organ-system
Safety of emetine assessed by rate of drug discontinuation | Up to 28 days
  Evaluate the safety of emetine assessed by rate of drug discontinuation

SECONDARY OUTCOMES:
Recovery (≥ 3 days without symptoms) | Up to 14 days
  Sustained resolution of all dengue symptoms for ≥ 3 consecutive days (where the first of those days is considered the date of recovery)
Time to Virologic Clearance of Dengue Virus by Qualitative RT-PCR | Pre-dose (day 0), day 3, and day 5
  Time to test negativity that is longitudinally measured by Qualitative real-time polymerase chain reaction (RT-PCR).
Quantitative Viral Load Assessment by RT-PCR Cycle Threshold (Ct) Values | Days 0,3, 5
  Measures of the average RT-PCR cycle threshold (Ct) values for dengue virus RNA at specified time points post-randomization.
Changes in inflammatory marker measured by hematocrit | Days 0 to 5
  Measure hematocrit in percentage (%) for patients
Changes in inflammatory marker measured by white blood count | Day 0-5
  Measure white blood count (WBC) for patients measured per microliter (mcL)
Changes in inflammatory marker measured by reticulocyte count | Day 0-5
  Measure reticulocyte count as percentage (%) for patients
Changes in inflammatory marker measured by platelet count | Day 0-5
  Measure platelet count for patients measured per microliter (mcL)
Changes in inflammatory marker measured by alanine aminotransferase | Day 0-5
  Measure alanine aminotransferase (ALT) for patients in units per liter (U/L)
Changes in inflammatory marker measured by serum bilirubin | Day 0-5
  Measure serum bilirubin for patients in milligrams per deciliter (mg/dL)
Changes in inflammatory marker measured by serum albumin | Day 0-5
  Measure serum albumin for patients in grams per deciliter (g/dL)
Changes in inflammatory marker measured by C-reactive protein | Day 0-5
  Measure C-reactive protein (CRP) for patients in milligrams per liter (mg/L)
Post infection fatigue measured by Fatigue Questionnaire | On Day 28
  Fatigue will be measured using the validated 11-item Fatigue Questionnaire (FQ), which assesses both physical (7 items) and mental (4 items) fatigue. Each item is rated on a 4-point Likert scale (0 = none, 3 = severe), with total scores ranging from 0 to 33, where higher scores indicate greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Kunchok Dorjee, MBBS, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Johns Hopkins University, Division of Infectious Disease, Baltimore, Maryland, United States
- Bharatpur Hospital, Bharatpur-10, Chitwan, Nepal

REFERENCES:
- [Background] Choy KT, Wong AY, Kaewpreedee P, Sia SF, Chen D, Hui KPY, Chu DKW, Chan MCW, Cheung PP, Huang X, Peiris M, Yen HL. Remdesivir, lopinavir, emetine, and homoharringtonine inhibit SARS-CoV-2 replication in vitro. Antiviral Res. 2020 Jun;178:104786. doi: 10.1016/j.antiviral.2020.104786. Epub 2020 Apr 3. PMID 32251767
- [Background] Ooi EE. Repurposing Ivermectin as an Anti-dengue Drug. Clin Infect Dis. 2021 May 18;72(10):e594-e595. doi: 10.1093/cid/ciaa1341. No abstract available. PMID 33124646
- [Background] Bhat CS, Shetty R, Sundaram B, Ramanan AV. Immunomodulatory therapy in dengue: need for clinical trials and evidence base. Arch Dis Child. 2023 Jun;108(6):451-452. doi: 10.1136/archdischild-2022-324100. Epub 2022 Jun 9. No abstract available. PMID 35680407
- [Background] Guzman MG, Gubler DJ, Izquierdo A, Martinez E, Halstead SB. Dengue infection. Nat Rev Dis Primers. 2016 Aug 18;2:16055. doi: 10.1038/nrdp.2016.55. PMID 27534439
- [Background] Beesetti H, Khanna N, Swaminathan S. Investigational drugs in early development for treating dengue infection. Expert Opin Investig Drugs. 2016 Sep;25(9):1059-69. doi: 10.1080/13543784.2016.1201063. Epub 2016 Jun 24. PMID 27322111
- [Background] Entner N, Grollman AP. Inhibition of protein synthesis: a mechanism of amebicide action of emetine and other structurally related compounds. J Protozool. 1973 Feb;20(1):160-3. doi: 10.1111/j.1550-7408.1973.tb06025.x. No abstract available. PMID 4347870
- [Background] Bleasel MD, Peterson GM. Emetine Is Not Ipecac: Considerations for Its Use as Treatment for SARS-CoV2. Pharmaceuticals (Basel). 2020 Nov 27;13(12):428. doi: 10.3390/ph13120428. PMID 33261173
- [Background] Grollman AP. Structural basis for inhibition of protein synthesis by emetine and cycloheximide based on an analogy between ipecac alkaloids and glutarimide antibiotics. Proc Natl Acad Sci U S A. 1966 Dec;56(6):1867-74. doi: 10.1073/pnas.56.6.1867. No abstract available. PMID 16591432